CLINICAL TRIAL: NCT00003118
Title: A Prospective Randomized Phase III Trial Comparing Trimodality Therapy (Cisplatin, 5-FU, Radiotherapy, and Surgery) to Surgery Alone for Esophageal Cancer
Brief Title: Surgery With or Without Chemotherapy and Radiation Therapy in Treating Patients With Cancer of the Esophagus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9781; U10CA031946 (NIH); CLB-C9781; E-C9781; NCCTG-C9781; RTOG-9716; CDR0000065873 (Registry Identifier: NCI Physician Desk Reference)
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Fluorouracil; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + Radiation + Surgery (Experimental)
  Interventions: Drug: cisplatin; Drug: fluorouracil; Procedure: surgical procedure; Radiation: radiation therapy
- Surgery (Active Comparator)
  Interventions: Procedure: surgical procedure

INTERVENTIONS:
Drug: cisplatin
  Arms: Chemotherapy + Radiation + Surgery
Drug: fluorouracil
  Arms: Chemotherapy + Radiation + Surgery
Procedure: surgical procedure
Radiation: radiation therapy
  Arms: Chemotherapy + Radiation + Surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether surgery is more effective with or without chemotherapy and radiation therapy for cancer of the esophagus.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without combination chemotherapy and radiation therapy in treating patients who have cancer of the esophagus that can be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall five-year survival rates and treatment failures in patients receiving neoadjuvant cisplatin (CDDP) plus fluorouracil (5-FU) with concomitant radiotherapy followed by surgical resection versus patients receiving surgery alone. II. Assess and compare the toxicities of each approach. III. Compare the incidence and pattern of local (gastric or esophageal bed or regional lymph nodes) and distant (supraclavicular lymph node, liver, peritoneal carcinomatosis, or lung, brain, etc.) recurrence. IV. Evaluate the prognostic ability of noninvasive and minimally invasive pretreatment staging with regard to survival and recurrence. V. Evaluate the ability of preresection adjuvant chemotherapy with concomitant radiation therapy to render tumors to lower stages. VI. Evaluate the impact of lymph nodes on survival and recurrence.

OUTLINE: This a two arm, randomized study. Patients are stratified by: cell type of cancer (squamous cell vs adenocarcinoma); lymph nodes (positive vs negative); and stage (invasive vs noninvasive). Patients in arm I undergo chemotherapy and radiotherapy within 24 hours of each other. Chemotherapy consists of cisplatin (CDDP) by bolus IV infusion over 30 minutes on day 1 and again on day 29. Fluorouracil (5-FU) is administered by continuous IV infusion for 4 days (on days 1-4 and 29-32) after completion of cisplatin. Radiotherapy is administered on days 1-5, 8-12, 15-19, 22-26, and 29-33, with a boost on days 36-38. If there is no disease progression or unresectable disease, surgery is performed within 3-8 weeks following completion of therapy. Patients in arm II undergo surgery alone no later than 6 weeks postrandomization. Patients are followed at least every 3 months for two years, then every 6 months for the next two years, and annually thereafter.

ELIGIBILITY:
1. Patients with histologically documented untreated squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (below 20 cm) or gastro-esophageal junction and with less than 2 cm distal spread into the gastric cardia were eligible.
2. No evidence of distant metastatic disease by history and physical examination
3. Upper endoscopy with biopsy, computed tomography (CT) of the chest and upper abdomen, and pulmonary function studies are required.
4. Bone scan is required for alkaline phosphatase more than 3X the institutional normal value.
5. Bronchoscopy is required if the primary tumor was adjacent to the trachea or left main stem bronchus.
6. Patients are required to have:

   * granulocyte counts ≥1,800/mL
   * platelet count ≥ 100,000/mL
   * creatinine clearance ≥ 50 mL/min
7. Esophageal ultrasound (EUS) and preresection staging by thoracoscopy (ts) and laparoscopy/minilaparotomy (ls), including biopsy of celiac axis and lesser curvature are recommended
8. Tumors must be considered surgically resectable (T1-3, NX), including regional thoracic lymph node (N1) metastases.
9. Patients with supraclavicular lymph nodes measuring ≤ 1.5 cm by CT (not palpable) are eligible.
10. Patients with lymph node metastases to levels 15 to 20 (predominantly celiac axis and paracardial nodes) ≤1.5 cm by CT.
11. Patients may not have previously received chemotherapy or radiation therapy for this tumor or any radiation therapy that would overlap the radiation fields required for this malignancy.
12. Patients with previous malignancies are eligible if more than 5 years had elapsed from diagnosis without evidence of tumor recurrence.
13. There can be no other serious illness that would limit survival to less than 2 years, or psychiatric condition that would prevent compliance with treatment or informed consent. Patients with uncontrolled or severe cardio- vascular disease,pulmonary disease, oractive infections are excluded.
14. Pregnant patients are excluded.
15. Informed consent is required for all patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1997-10; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Krasna, MD, Study Chair — Jersey Shore University Medical Center
Locations (38):
- United States (38):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Result] Krasna M, Tepper JE, Niedzwiecki D, et al.: Trimodality therapy is superior to surgery alone in esophageal cancer: results of CALGB 9781. [Abstract] American Society of Clinical Oncology 2006 Gastrointestinal Cancers Symposium, 26-28 January 2006, San Francisco, California. A-4, 2006.
- [Result] Tepper JE, Krasna M, Niedzwiecki D, et al.: Superiority of trimodality therapy to surgery alone in esophageal cancer: results of CALGB 9781. [Abstract] J Clin Oncol 24 (Suppl 18): A-4012, 2006.